CLINICAL TRIAL: NCT04386200
Title: Educational Approach, Clinical Nutrition and Type 2 Diabetes: Traditional Strategies and Innovative Technologies
Brief Title: Web-based Approach in Nutrition and Diabetes
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Università degli Studi 'G. d'Annunzio' Chieti e Pescara (Other)
Responsible Party: Principal Investigator, Ester Vitacolonna, Professor, Università degli Studi 'G. d'Annunzio' Chieti e Pescara
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VITA02
Record Dates: First submitted 2020-05-05; First posted 2020-05-13 (Actual); Last update posted 2020-05-15 (Actual); Status verified 2020-05

CONDITIONS: Type 2 Diabetes Mellitus; Overweight and Obesity; Nutritional and Metabolic Diseases
Keywords: Web technologies; Nutrition
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Overweight; Obesity; Nutritional and Metabolic Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WEB GROUP (Experimental): Traditional approach integrated with web-based technologies.
  Interventions: Other: web-based thecnologies
- TRADITIONAL GROUP (Other): Traditional educational approach
  Interventions: Behavioral: traditional approach

INTERVENTIONS:
Other: web-based thecnologies — Integration of "traditional" face-to-face educational approach with web-based technologies.
  Arms: WEB GROUP
Behavioral: traditional approach — "traditional" face-to-face educational approach
  Arms: TRADITIONAL GROUP

SUMMARY:
The study aims to test web-based strategies, in overweight or obese participants at risk or affected by Type 2 Diabetes Mellitus , to promote adherence over time to a healthy lifestyle and nutritional medical therapy (TMN). The study population includes 40 subjects, randomly allocated to web group (therapeutic reinforcement through web-based strategies) or traditional group (traditional educational approach). Anthropometric and clinical parameters will be collected, as well as scores of validated questionnaires will be administered up to 12 months from the enrollment.

ELIGIBILITY:
Inclusion Criteria:

* Overweight or obesity (BMI ≥25 kg/m2)
* Participants with or at risk of Type 2 Diabetes Mellitus
* Skills in the use web-based technologies and internet accessibility

Exclusion Criteria:

* Conditions that could interfere with the execution and completion of the project or failure adherence to the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2019-02-13 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Body Weight | Baseline, month 3, month 6, month 9 and month12
  Assessment of body weight (in kilograms) at baseline and after 3, 6, 9 and 12 months

SECONDARY OUTCOMES:
Change from baseline in BMI | Baseline, month 3, month 6, month 9 and month12
  Assessment of BMI (kg/m^2) at baseline and after 3, 6, 9 and 12 months
Change from baseline in body circumferences | Baseline, month 3, month 6, month 9 and month12
  Assessment of body circumferences (in centimeters) at baseline and after 3, 6, 9 and 12 months
Change from baseline in Systolic and Diastolic blood pressure | Baseline, month 3, month 6, month 9 and month12
  Assessment of Systolic and Diastolic blood pressure (mm hg) at baseline and after 3, 6, 9 and 12 months
Change from baseline in fasting blood glucose | Baseline, month 3, month 6, month 9 and month12
  Assessment of fasting blood glucose (mg/dl) at baseline and after 3, 6, 9 and 12 months
Change from baseline in HbA1C | Baseline, month 3, month 6, month 9 and month12
  Assessment of HbA1C at baseline and after 3, 6, 9 and 12 months
Change from baseline in Dietary habits estimated by PREvencion con DIetaMEDiterranea questionnaire (PREDIMED questionnaire) | Baseline, month 3, month 6, month 9 and month12
  Assessment of Dietary habits at baseline and after 3, 6, 9 and 12 months. Changes in dietary habits will be estimated using a 14-item PREDIMED questionnaire which is a questionnaire to assess the adherence to the Mediterranean diet, 0 being the minimum total score and 14 the maximum total score. Higher values represent a higher adherence to the Mediterranean diet.
Change from baseline in physical activity level estimated by the International Physical Activity Questionnaire (IPAQ) - short form | Baseline, month 3, month 6, month 9 and month12
  Assessment of physical activity level at baseline and after 3, 6, 9 and 12 months. Changes in the level of physical exercise will be estimated by the International Physical Activity Questionnaire (IPAQ-short form) which is a questionnaire to assess the level of physical activity. Patients are asked to measure the average amount of time spent in sedentary behaviours and different intensity levels of physical activity. The questionnaire obtains three different intensity levels of physical activity: low, moderate and high.
Change from baseline in Quality of life by 36-item short form health survey (SF-36) | Baseline, month 3, month 6, month 9 and month12
  Assessment of Quality of life by SF-36 at baseline and after 3, 6, 9 and 12 months. The 36-Item Short Form Health Survey (SF-36) is a self-report generic quality of life measure. The SF-36 measures eight scales: physical functioning (PF), role physical (RP), bodily pain (BP), general health (GH), vitality (VT), social functioning (SF), role emotional (RE), and mental health (MH) with scores ranging from 0 to 100. Higher scores indicate greater self-reported quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital "SS Annunziata", Chieti, Italy

REFERENCES:
- [Derived] Fraticelli F, Nicola MD, Vitacolonna E. A nutritional web-based approach in obesity and diabetes before and during the COVID-19 lockdown. J Telemed Telecare. 2023 Feb;29(2):91-102. doi: 10.1177/1357633X20966933. Epub 2020 Oct 21. PMID 33081596